CLINICAL TRIAL: NCT05337917
Title: Long-term Hand Function and Sensation Following Digital Nerve Injury and Repair- a Case Control Study.
Brief Title: Digital Nerve Injury - a Case Control Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, Principal investigator, Karolinska Institutet
Other Study IDs: Digital nerve clinical results
Record Dates: First submitted 2022-01-29; First posted 2022-04-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Digital Nerve Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Injury to digital nerve: thumb, digit II radial side, digit V ulnar side
  Interventions: Procedure: Surgical of the digital nerve
- Control: Injury to digital nerve: digit II ulnarside, dig III, dig IV dig V radial side.
  Interventions: Procedure: Surgical of the digital nerve

INTERVENTIONS:
Procedure: Surgical of the digital nerve — All patients (cases and controls) were subject to surgical repair of digital nerve injury.

SUMMARY:
Case control study, investigating what hand function and sensory function do patients perform 3-10 years following digital nerve injury and repair. The aim is to investigate if hand function is more limited following digital nerve injury in the thumb, index- and little finger, compared to less unburdened sensory surfaces in the fingers. Secondary aim is to investigate the long term sensory function following digital nerve injury.

DETAILED DESCRIPTION:
Eligible patients are individuals treated at the Department of Hand surgery in Stockholm, Sweden during 2012-2018. Inclusion criteria include diagnostic codes (ICD-10) for a digital nerve injury in the thumb (S64.3) or finger (S64.4) in combination with the surgical code (KKÅ97) Nomesco classification of surgical procedures for nerve repair (ACB29). Exclusion criteria are concomitant flexor tendon injury and/or skeletal injury, amputations, and severe soft tissue injuries. Patients residing outside the Stockholm region and children below 18 years of age are also excluded. Initially a total number of 1330 patients have been identified. All medical records have been thoroughly scrutinized. After excluding concomitant tendon injury, a total of 606 patients remained with isolated digital nerve injury. A randomly selected sample of participants have been assigned to two groups: Patients with an injury to the digital nerve of the thumb, digit II radial side, digit V ulnar side were assigned to the "case" group and matched "controls" were randomly selected among patients with an injury to the digital nerves of either the ulnar side of digit II, either nerve of digit III and digit IV or the radial nerve of digit V. Cases and controls have been matched according to sex, year of injury and patient age.

For the purpose of this study, a clinical evaluation to investigate hand function, sensory function, strength, and ability to discriminate warm and cold and sharp and dull will be conducted. Questionnaires are used for Patient Reported Outcome Measures (PROM): Disability of the Arm Shoulder, and Hand (QuickDASH), Patient questionnaire HQ8 arm and hand (HQ8), The Hospital Anxiety and Depression Scale (HADS), Saltin-Grimby Physical Activity Level Scale (SGPALS), and in addition Douleur Neuropathique en 4 Questions (DN4) for assessment of neuropathic pain will be performed. All outcomes will be compared between groups defined as case (digital injury to the thumb, radial nerve of the index finger or ulnar nerve of the little finger) or control (all other digital nerve injuries).

ELIGIBILITY:
Inclusion Criteria:

* diagnostic codes (ICD-10) for a digital nerve injury in the thumb (S64.3) or finger (S64.4) in combination with the surgical code (KKÅ97) Nomesco classification of surgical procedures for nerve repair (ACB29).
* treatment completed in Södersjukhuset hospital 2012 - 2018

Exclusion Criteria:

* concomitant skeletal injury,
* amputations
* severe soft tissue injuries
* microvascular reconstruction
* residence outside the Stockholm region
* patient age below 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with digital nerve injury were identified from a registry cohort consisting in 1330 patients. They were all treated due to a digital nerve injury at our hospital 2012 - 2018. A random sample of cases and controls were selected, matched for time from injury to evaluation, age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Handfunction | 3-10 years post operatively
  Measured by Mini Sollerman test for handfunction.

SECONDARY OUTCOMES:
Sensation | 3-10 years post operatively
  Semmes Weinstein, Static two point discrimination
Sensation | 3-10 years post operatively
  Static two point discrimination
Patient Rated Outcome Measure (PROM) for hand function | 3-10 yrs post op
  QuickDASH (Disability of the Arm Shoulder and Hand)
PROM for hand function | 3-10 yrs post op
  HQ8 (HAKIR Questionnaire 8 questions)
PROM for hand function | 3-10 yrs post op
  SGPALS (Saltin-Grimby Physical Activity Level Scale)
PROM for neuropathic pain | 3-10 yrs post op
  DN4 (Douleur neuropathique 4 levels)
PROM for depression and anxiety | 3-10 yrs post op
  HADS (Hospital Anxiety and Depression Scale)
PROM | 3-10 yrs post op
  Physical activity scale.
Range of motion | 3-10 yrs post op
  Goniometer measurements of finger joints
Pinch strength | 3-10 yrs post op
  Grip strength as measured by Pinch gauge
Strength | 3-10 yrs post op
  Grip strength as measured by JAMAR

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Mellstrand Navarro, MD Prof, Principal Investigator — Region Stockholm
Locations (1):
- Linda Evertsson, Stockholm, Sweden